CLINICAL TRIAL: NCT02339051
Title: The Effect of Mechanical Loading on Bone Material Strength and Microarchitecture in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mattias Lorentzon (Other)
Responsible Party: Sponsor-Investigator, Mattias Lorentzon, Professor, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 563-14
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Osteoporosis; Postmenopause
Keywords: Basic Science
MeSH Terms: conditions — Osteoporosis

ARMS (1):
- One leg jumping (Experimental): Study subjects will jump on one leg on repeated occasions (incremental daily repetitions) for a period of three months. The same leg will be used for jumping throughout the study. The other leg will serve as control.
  Interventions: Behavioral: Jumping on one leg

INTERVENTIONS:
Behavioral: Jumping on one leg

SUMMARY:
Osteoporosis is a large public health disease, characterized by low bone mass and micro architectural deterioration of bone tissue, resulting in enhanced bone fragility and consequent increase in fracture risk. Osteoporosis is present when bone mineral density (BMD) or content (BMC), measured by dual-energy X-ray absorptiometry (DXA), is more than 2.5 SDs below the mean value of the young adult. BMD measured by DXA is a surrogate measure of bone strength and is the primary determinant of fracture risk in both men and women. However, the majority of fragility fractures occur in women and in individuals who do not have osteoporosis according to these standards, indicating that BMD is just one among several indicators of bone health and that assessment of fracture risk should also rely on other bone properties. Newer imaging methods, such as quantitative computerized tomography (QCT), can complement information from DXA-measurements due to its ability to assess volumetric BMD and bone geometry and to differentiate between cortical and trabecular bone compartments. Bones are composite materials made predominantly of living cells, extracellular matrix, water and lipids. This composite nature of the bone material enables it to absorb stresses by elastic deformation and to endure high loads before fracturing. A new in vivo measurements of bone material strength can be used to evaluate bone mechanical properties and thereby the fracture risk. It is well established that the skeleton benefits, in terms of increased density, from regular physical activity. However, changes in BMD are still the main surrogate for assessing improvements in exercise-induced bone health despite the experimental findings as well as findings in humans showing that improvements in mechanical bone properties are independent of changes in BMD. These improvements in mechanical bone properties may be due to changes in bone shape or matrix composition. It could then be argued that a decrease in BMD is only one of the possible manifestations of osteoporosis and that bone strength or fragility is multifactorial. The objective for this study is to investigate the role of mechanical loading on bone material strength and bone microarchitecture in middle-aged women. The overall hypothesis is that mechanical loading is a regulator of bone material strength and microarchitecture in middle-aged women. This is an intervention study where the participants will act as their own controls. The investigators intend to include 40 postmenopausal and healthy women 50-60 years of age in the study. Advertisements in local papers and at the hospital will be used to come into contact with suitable study subjects. The women will be asked to perform an intervention program, including jumping on one leg every day during a 3-month period according to a protocol with a gradually increasing load/number of jumps. The women have to choose one of their legs as intervention-leg and stick to the chosen leg throughout the study. The leg without intervention will be used as a control. Both bone material strength (BMS) and bone microarchitecture will be measured before and after intervention in both legs (tibia). The operators measuring BMS (OsteoProbe®) and bone microarchitecture (high resolution pQCT) will be blinded concerning each participant's choice of leg for intervention. In addition, subjects will be asked to register daily physical activity in a structured diary. The primary outcome measure will be changes in bone material strength (BMS) in the lower leg (tibia) with intervention compared to the leg (tibia) without intervention. Participants will attend two clinic visits, at baseline and after 3 months when the intervention period is completed. The secondary outcome measures will be changes in total volumetric density, cortical volumetric density, cortical cross sectional area and trabecular bone volume fraction in the lower leg (tibia) with intervention compared to the leg (tibia) without intervention.

ELIGIBILITY:
Inclusion Criteria:

* aged between 50 and 60 years,
* no history of osteoporosis,
* not undertaken resistance training and/or weight-bearing impact exercise more than once a week in the past three months,
* be able and willing to perform the intervention program (one leg jumping), and
* be reachable via telephone once weekly throughout the study

Exclusion Criteria:

* current smoking,
* current or prior (past 6 months) use of hormone replacement therapy,
* having sustained a low trauma fragility fracture in the past 6 months,
* any medical condition (e.g. type 1 diabetes,
* chronic kidney failure or liver disease, cancer) or
* use of medication known to influence bone metabolism or fracture risk (e.g. glucocorticoids, thiazide diuretics, anticonvulsants, bisphosphonates), or
* initiating calcium or vitamin D supplementation in the preceding 6 months

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Changes in bone material strength in the tibia (measured using OsteoProbe®) | Three months
  Bone material strength measured using OsteoProbe®

SECONDARY OUTCOMES:
Changes in total volumetric density in the tibia (Measured using high-resolution pQCT device (HR-pQCT) | Three months
  Measured using high-resolution pQCT device (HR-pQCT) (XtremeCT, Scanco Medical AG, Switzerland)
Changes in cortical volumetric density in the tibia (Measured using high-resolution pQCT device (HR-pQCT) | Three months
  Measured using high-resolution pQCT device (HR-pQCT) (XtremeCT, Scanco Medical AG, Switzerland)
Changes in cortical cross sectional area in the tibia (Measured using high-resolution pQCT device (HR-pQCT) | Three months
  Measured using high-resolution pQCT device (HR-pQCT) (XtremeCT, Scanco Medical AG, Switzerland)
Changes in trabecular bone volume fraction in the tibia (Measured using high-resolution pQCT device (HR-pQCT) | Three months
  Measured using high-resolution pQCT device (HR-pQCT) (XtremeCT, Scanco Medical AG, Switzerland)